CLINICAL TRIAL: NCT05528783
Title: Application of FIT-DNA Detection in Following Colorectal Cancer Resection-Implications for Surveillance
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: New Horizon Health (Unknown)
Responsible Party: Principal Investigator, ZHI-ZHONG PAN, Professor, Director, M.D., Ph.D, Sun Yat-sen University
Other Study IDs: 2021-AFFCCR
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; FIT-DNA; Detection
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer (CRC) is a common cancer that threatens human health, with the incidence ranking the third in the world. 70% of patients are in the middle and late stages whendiagnosed, and even after radical surgery, 30% - 50% of patients with CRC have recurrence or metastasis after radical surgery. Therefore, after radical surgery and adjuvant chemotherapy, regular monitoring of CRC patients should be paid attention to in order to detect the recurrence and metastasis lesions that can be resected and the early non-invasive metachronous multiple primary tumors.

The sensitivity of FIT-DNA to CRC was 95.5%, the sensitivity to advanced adenoma (AA) was 63.5%, and the specificity was 87.5%, showing a good ability to screen colorectal cancer and precancerous lesions.

At present, there is no report on the application of FIT-DNA combined detection technology in the high-risk recurrence period and mid - and long-term monitoring after CRC surgery in China. In this study, Fit-DNA combined detection technology was applied to the follow-up monitoring of patients after CRC surgery, so as to optimize the current typical postoperative follow-up strategy, find early recurrence and multiple primary colorectal tumors after CRC surgery, seek the best postoperative follow-up model, improve the compliance of patients to follow-up, and ultimately benefit survival.

Detailed Description:Outline:This study was a single-center, observational study. Fit-DNA detection technology was used as a target method, and colonoscopy was used as the gold standard control to follow up and monitor patients with colorectal tumors after surgery, and to explore whether it is an effective non-invasive auxiliary method for monitoring CRC recurrence and metastasis and multiple primary colorectal tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1). The pathological diagnosis was colorectal adenocarcinoma； 2). Age: 18 to 80 years old,allgenders； 3). Radical surgery for CRC is required； 4). No preoperative antitumor therapy (including chemotherapy, radiation therapy, targeted therapy, and immunotherapy)； 5). Preoperative examination revealed no distant metastasis； 6). There were no severe hemorrhoids or other known conditions that can cause gastrointestinal bleeding before surgery； 7). The clinical treatment data were complete；

Exclusion Criteria:

* 1). With a history of digestive tract tumors other than CRC； 2). Previous colorectal surgery； 3). Patients requiring a fistula； 4). With complete intestinal obstruction or perforation； 5). Women who are pregnant or breastfeeding； 6). Patients with metastases found in other sites during surgery that cannot be removed radically； 7). Patients unwilling or unable to sign an informed consent form； 8). A strict vegetarian； 9). Patients who are unwilling to follow up according to the protocol or have poor follow-up compliance； 10). Any conditions that the study physician deemed inappropriate for inclusion。

Exit or terminate criteria：

1. . Follow-up information for the patients was not available
2. . Distant metastasis was diagnosed after surgery
3. . Subjects died before the end of follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were newly diagnosed with colorectal cancer by colorectal endoscopy and required surgical radical surgery for TNM stage I, II and III non-stoma patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic sensitivity and specificity of FIT-DNA detection for local recurrence and advanced colorectal neoplasm of CRC. | up to 5 years
  The diagnostic sensitivity and specificity of FIT-DNA detection for local recurrence and advanced colorectal neoplasm of CRC.

SECONDARY OUTCOMES:
1.The AUC of FIT-DNA in recurrent CRC and advanced colorectal stage. | up to 5 years
  1.The AUC of FIT-DNA in recurrent CRC and advanced colorectal stage.
2.NPV、PPVof FIT-DNA in recurrent CRC and advanced colorectal stage. | up to 5 years
  2.NPV、PPVof FIT-DNA in recurrent CRC and advanced colorectal stage.
3.The time interval between CRC recurrence and advanced colorectal neogenesis after the first positive appearance was detected by FIT-DNA detection. | up to 5 years
  3.The time interval between CRC recurrence and advanced colorectal neogenesis after the first positive appearance was detected by FIT-DNA detection.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorectal Department,SunYat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Share to New Horizon Health